CLINICAL TRIAL: NCT06343571
Title: Longitudinal Outcomes in MED-EL Cochlear Implant Recipients Using a FLEX Electrode Array: a Retrospective Study
Brief Title: Longitudinal Outcomes in MED-EL Cochlear Implant Recipients Using a FLEX Electrode
Acronym: LOTOS
Status: Completed | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EL_CRD_2022_12
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cochlear Implants
Keywords: cochlear implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims at analysing data from clinical routine as anonymized data sets. The study aims at analysing clinical data from MED-EL Cochlear Implant (CI) recipients using a FLEX electrode array.

ELIGIBILITY:
Inclusion Criteria:

* MED-EL CI recipients
* FLEX electrode array

Exclusion Criteria:

* Lack of compliance with any inclusion criterion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There is no requirement to actively participate in the study for any of the subjects.
  This study consists of a one-time data extraction from a clinical database. Data will be included from 03/2006 to date of extraction
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Evaluate short and long term longitudinal clinical performance data from MED-EL CIs to assess their clinical effectiveness and safety. | Through study completion: single data extraction (3 month to completion)
  Longitudinal data from clinical routine

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Büchner, Prof, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No